CLINICAL TRIAL: NCT06410092
Title: A Phase 1, First-in-Human, Open-Label, Dose Escalation and Dose Expansion Study of FTL001 in Patients With Advanced or Metastatic Solid Tumors
Brief Title: Study in Patients With Advanced Solid Malignancies to Evaluate the Safety of FTL001
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Sound Biopharmaceuticals Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: FTL001-101
Record Dates: First submitted 2024-04-30; First posted 2024-05-10 (Actual); Last update posted 2024-05-10 (Actual); Status verified 2024-05

CONDITIONS: Solid Tumor
Keywords: Solid Tumor; FTL001; Sound Biopharmaceuticals

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Arm 1 Part 1 Dose Escalation (Experimental): Escalating doses of FTL001 depending on cohort at enrollment
  Interventions: Drug: FTL001
- Arm 1 Part 2 Dose Expansion (Experimental): Two dose groups of FTL001 depending on data of Arm 1 Part 1
  Interventions: Drug: FTL001

INTERVENTIONS:
Drug: FTL001 — IV infusion every 2 weeks

SUMMARY:
This is an open, multi-center, Phase I clinical study to evaluate the safety, tolerability, pharmacokinetics/pharmacokinetics and initial efficacy of FTL001 in patients with advanced and metastatic solid tumors.

DETAILED DESCRIPTION:
The study is divided into two phases, Part 1 (FTL001 dose escalation) and Part 2 (FTL001 dose expansion), and is intended to include approximately 26-44 participants.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must give informed consent to this study prior to the study and sign a written informed consent form voluntarily;
2. Age ≥18 and ≤75, both male and female;
3. Expected survival time of more than 3 months;
4. Histologically or cytologically confirmed advanced solid tumors;
5. Patients with advanced recurrence, metastasis and refractory solid tumors whose disease progresses after standard treatment or who are intolerant to standard treatment or have no standard treatment (the definitions of standard treatment and refractory recurrence refer to authoritative diagnosis and treatment guidelines at home and abroad);
6. At least 1 measurable lesion at baseline according to the definition of RECISTv1.1;
7. ECOG performance score of 0 or 1;
8. Adequate organ function;
9. Fertile men or women with the possibility of becoming pregnant, using an effective contraceptive method during the trial, and continuing contraception for 6 months after the end of treatment;

Exclusion Criteria:

1. Have a history of malignancies other than the disease studied within the previous 5 years, except for malignancies that have been cured after treatment and have no risk of recurrence (including but not limited to adequately treated thyroid cancer, cervical carcinoma in situ, basal or squamous cell skin cancer, or breast ductal carcinoma in situ treated with radical surgery);
2. Prior anticancer therapy (chemotherapy, targeted agents, radiotherapy, and immunotherapy) within 28 days before first dose;
3. Prior treatment with any anti-CD137 antibody or drug (single agent or combination);
4. Adverse reactions caused by previous treatment that did not recover to CTCAE (version 5.0) grade 1 or below, hair loss, neurotoxicity to CTCAE (version 5.0) grade 2 or below, or other adverse reactions that researchers judged to have no safety risk could be included;
5. Previously received allogeneic hematopoietic stem cell transplantation or solid organ transplantation;
6. Active primary or metastatic tumors of the central nervous system (except in patients who have previously been treated and discontinued treatment 4 weeks before the first study drug administration, symptomless patients who do not require long-term glucocorticoid therapy), seizures, spinal cord compression, or carcinomatous meningitis;
7. Have or have suspected active autoimmune diseases, including but not limited to systemic lupus erythematosus, rheumatoid arthritis, inflammatory bowel disease, etc., but the following conditions can be included: Type 1 diabetes that can be controlled by alternative therapy alone, skin diseases that do not require systemic treatment (e.g. Psoriasis, vitiligo);
8. Suffering from clinical symptoms or symptomatic treatment of pleural fluid or ascites;
9. Severe cardiovascular and cerebrovascular diseases, such as uncontrolled or poorly controlled high blood pressure or Pulmonary hypertension; Unstable angina pectoris or myocardial infarction, coronary artery bypass grafting or stenting within 6 months prior to study administration; Chronic heart failure with heart function ≥2 (NYHA rating); Degree II and above heart block; Left ventricular ejection fraction (LVEF) < 50%; Study cerebrovascular accident (CVA) or transient ischemic attack (TIA) within 6 months prior to medication;
10. History of pulmonary disease: interstitial pneumonia, obstructive pulmonary disease and symptomatic bronchospasm;
11. Active infection requiring intravenous anti-infective treatment, or unhealed wounds or ulcers occurring within 14 days prior to initial administration;
12. Test positive for human immunodeficiency virus (HIV) antibodies;
13. Hepatitis (non-alcoholic steatohepatitis, alcoholic or drug-related, autoimmune hepatitis) and cirrhosis with portal hypertension; Active hepatitis B or C:
14. Active tuberculosis (TB) is known to exist. Subjects suspected of active TB should be examined for chest X-rays, sputum, and clinical signs and symptoms.
15. Received systemic corticosteroids (prednisone > 10 mg/ day or equivalent) or other immunosuppressive drugs within 14 days prior to the initial study;
16. Receive live vaccination within 4 weeks prior to the initial study administration;
17. Major surgical procedures within 4 weeks prior to initial study medication (as defined by the investigator, open biopsy, severe trauma, etc.). Note: It is acceptable to replace an intravenous drip dropper. Had a major surgical procedure planned within 30 days of initial dosing (as determined by the investigator). Local procedures (such as placement of systemic ports, air-core needle biopsies, and prostate biopsies) are permitted, provided that the procedure is completed at least 24 hours before the first administration of the investigational therapeutic agent;
18. Pregnant or lactating women;
19. History of hypersensitivity or idiosyncrasy to the excipients of the study drug or to any monoclonal antibody;
20. Those who have previously received cellular immunotherapy (CAR-T).

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 44 (Estimated)
Dates: Start 2023-06-05 (Actual); Primary Completion 2026-01 (Estimated); Study Completion 2027-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants with dose-limiting toxicities (DLTs) | First Cycle (28 days)
  Number of participants with DLTs during the 28 days following the first administration of FTL001

SECONDARY OUTCOMES:
To preliminarily evaluate the anti-tumor activity | every 2 cycles (each cycle is 28 days)
  Computed tomography (CT) scans of tumors will be evaluated according to RECIST 1.1 and iRECIST (2017).
Pharmacokinetic (PK) measure: Maximum observed serum concentration (Cmax) | From first dose (Cycle 1 Day 1, each cycle is 28 days) until the last dose (up to 2 years)
  PK samples will be collected at predefined timepoints to determine Cmax.
Pharmacokinetic (PK) measure: Area under the plasma concentration versus time curve (AUC) | From first dose (Cycle 1 Day 1, each cycle is 28 days) until the last dose (up to 2 years)
  PK samples will be collected at predefined timepoints to determine AUC.

CONTACTS AND LOCATIONS:
Overall Officials: Yuankai Shi, MD, Principal Investigator — Cancer Institute and Hospital, Chinese Academy of Medical Sciences; Shoubin Wen, MD, Study Director — Sound Biopharmaceuticals Ltd.
Locations (3):
- China (3):
  - Cancer Institute and Hospital, Chinese Academy of Medical Sciences, Beijing, Beijing Municipality
  - Chongqing University Cancer Hospital, Chongqing, Chongqing Municipality
  - West China Hospital, Chengdu, Sichuan

IPD SHARING:
Plan to Share IPD: No